CLINICAL TRIAL: NCT02643654
Title: A Double-blind, Randomised, Placebo-controlled Clinical Trial of the Efficacy of MABp1, a- First-in-class True Human Antibody Targeting Interleukin-1alpha, in Patients With Hidradenitis Suppurativa Not Eligible for antiTNF Therapy
Brief Title: MABp1 IN HIDRADENITIS SUPPURATIVA REFRACTORY TO ADALIMUMAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evangelos J. Giamarellos-Bourboulis, M.D. (Other)
Collaborators: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor-Investigator, Evangelos J. Giamarellos-Bourboulis, M.D., Associate Professor of Internal Medicine, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIDRA04
Record Dates: First submitted 2015-12-20; First posted 2015-12-31 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: interleukin-1alpha
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo product is manufactured following the same procedures and batch records used to manufacture the MABp1 drug product. The placebo dosage form is a sterile isotonic formulation buffer at pH 6.2-6.5. Each 10-ml Type I borosilicate glass serum vial contains 6mL of the formulation buffer, and is sealed with a 20-mm Daikyo Flurotec butyl rubber stopper and flip-off aluminum seal.
  Interventions: Drug: Placebo
- MABp1 (Active Comparator): MABp1 is a recombinant human IgG1 monoclonal antibody specific for human interleukin-1α (IL-1α). The entire MABp1 heavy and light chain sequences are identical to those found in naturally-occurring human IgG1κ, with the light and heavy chain variable regions being identical to those originally expressed by a peripheral blood B lymphocyte that was obtained from a healthy individual. It is a sterile injectable liquid formulation of 50 mg/mL MABp1 in a stabilizing isotonic buffer (pH 6.4). Each 10-mL serum vial contains 6 ml of the formulation, and is sealed with a 20-mm grey bromobutyl stopper and flip-off aluminum seal
  Interventions: Drug: MABp1

INTERVENTIONS:
Drug: MABp1 — This is a sterile injectable liquid formulation of 50 mg/mL MABp1 in a stabilizing isotonic buffer (pH 6.4). Each 10-mL serum vial contains 6 ml of the formulation, and is sealed with a 20-mm grey bromobutyl stopper and flip-off aluminum seal
  Arms: MABp1
Drug: Placebo — The placebo dosage form is a sterile isotonic formulation buffer at pH 6.2-6.5. Each 10-ml Type I borosilicate glass serum vial contains 6mL of the formulation buffer, and is sealed with a 20-mm Daikyo Flurotec butyl rubber stopper and flip-off aluminum seal.
  Arms: Placebo

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic inflammatory skin disorder. Although adalimumab is recently licensed for moderate to severe HS, many cases fail to respond or relapse during treatment. Favorable outcomes from a recently conducted double-blind randomized clinical study on the efficacy of anakinra, one interleukin(IL)-1alpha blocker, in hidradenitis suppurativa (HS), led to validate the efficacy of MABp1, a true human antiIL-1α antibody in these cases.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic devastating skin disorder affecting areas rich in apocrine glands. Nodules appear in the affected areas; they progressively become swollen and rupture with the release of pus. This process occurs repeatedly leading to sinus tract formation and scars. This disease course creates a frustrating situation not only for the patients but also for physicians. Traditional treatments comprise short-courses of antibiotics and surgical excision. However, relapse is the rule so that HS leads to severe impairment of the quality of life. The Dermatology Quality Life Index (DQLI) for HS is 8.9, being higher than any other skin disorder.

This devastating disorder has often been neglected and considered a rare situation. However, HS seems to indiscriminately affect the global population. A large epidemiological survey in France reports 0.97% disease prevalence.

The exact pathophysiology of HS is unknown. Both familial and non-familial cases of HS exist. Familial HS is less than 5% of cases and it is usually inherited through the dominant autosomal mode. Mutations in genes encoding for the gene complex of nicastrin-γ-secretase are predominant in hereditary HS. However, little is known on the genetic predisposition of non-familial HS that comprises the great majority of cases. Two studies by the investigators have been conducted to explore the predisposition of HS among patients who carry single nucleotide polymorphisms (SNPs) of gene encoding for pro-inflammatory cytokines namely TNF and IL-12RB1. Results have shown that carriage of haplotypes comprising minor frequency SNP alleles at the promoter region of TNF increases the likelihood for HS; furthermore these patients are less likely to respond to treatment with anti-TNF agents. In parallel, haplotyping for gene SNPs of exon 7 and exon 10 of IL-12RB1 comprising seven constitutive SNPs has shown that carriage of the h2 haplotype composed by four minor frequency SNP alleles is associated with more severe disease phenotypes. These results indicate a strong component of the implication of the innate immune responses in the pathogenesis of HS. In conjunction with this and following a successful phase II trial, the two phase III PIONEER studies ended up with significant improvement of patients after 12 weeks of treatment with adalimumab. A novel score, HS clinical response (HiSCR) score, was introduced in these trials and it is now suggested for the evaluation of the efficacy of any new formulation in HS. Using this score, it was found that the success rate of adalimumab to achieve a positive HiSCR after 12 weeks of treatment ranged between 40 and 60%. This means that several patients do not respond to adalimumab treatment whereas others may relapse after some initial response.

The investigators have recently concluded a phase 2, double-blind, randomized study of the efficacy of anakinra treatment administered 100mg subcutaneously daily for 12 consecutive weeks compared to placebo in 19 patients; 10 were allocated to the placebo arm and nine to the anakinra arm (EudraCT2011-005145-12, www.clinicaltrials.gov NCT01558375). Results were favorable for the clinical efficacy of anakinra. The primary endpoint defined to be disease activity was marginally achieved in the modified intent-to-treat population. Regarding the secondary endpoints, treatment with anakinra was very effective in: a) prolonging the time to new exacerbation compared to the placebo arm; and b) modulating cytokine stimulation from peripheral blood mononuclear cells. More precisely, the production of interferon-γ was significantly decreased and the production of IL-22 was increased compared to the placebo arm. HiSCR score was not initially included as a study endpoint because this score has not been developed when the trial was submitted to the authorities. Retrospective validation of the HiSCR score showed significant reduction at week 12 in 7 patients (77.8%) treated with anakinra compared to three patients (30%) treated with placebo (p: 0.039).

The considerable efficacy of anakinra that blocks interleukin (IL)-1alpha (IL-1α) leads to consider a significant role of IL-1α in the pathogenesis of HS. MABp1 is a first-in-class true human monoclonal antibody cloned directly from a human B lymphocyte and specifically targets IL-1α. Results from a first-in-man trial were recently published, in which fifty-two patients with metastatic cancer were enrolled in an open-label phase 1 study. The drug was well-tolerated, tumor responses were observed, and interestingly, treatment was accompanied by an increase of lean body weight.

The purpose of this clinical study is to evaluate the safety and the efficacy of MABp1 compared to placebo in patients with moderate to severe HS who either failed previous treatment with antiTNF regimens or who relapsed under antiTNF regimens or who are treatment naïve and they are unwilling to receive subcutaneous adalimumab treatment. The rationale behind the promising success of MABp1 relies on recent findings showing heterogeneity of cytokines in skin lesions with several patients expressing huge concentrations of TNFα the lesions and other who express low concentrations of TNFα but huge concentrations of IL-1α.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the patient
* Age equal to or more than 18 years
* Diagnosis of hidradenitis suppurativa (HS)
* HS of Hurley II or III stage disease or rapidly progressive HS of Hurley I stage
* Presence of at least 3 inflamed nodules consistent with HS in the body
* At least one of the following: a) previous failure of treatment with any anti-TNF regimen; b) previous relapse under treatment with any anti-TNF regimen; c) unwillingness to receive subcutaneous adalimumab treatment

Note: Since rapidly progressive HS of Hurley I stage as defined below is not a licensed indication for adalimumab, these patients can be enrolled irrespective or not of a history of previous adalimumab treatment.

Exclusion Criteria:

* History of systemic lupus erythematosus
* Treatment with any biologicals or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies.
* Administration of any live (attenuated) vaccine over the last 4 weeks
* History of recurrent vein thrombosis or embolism compatible with anti-cardiolipin syndrome
* Any present serious bacterial infection namely pneumonia, endocarditis, acute pyelonephritis and intrabdominal infection. These patients can be enrolled once the attending physicians confirm cure by the infection
* Hepatic dysfunction defined as any value of transaminases, of γ-glutamyl transpeptidase or of bilirubin> 2 x upper normal limit
* History of haematological or solid tumor malignancy, arterial hypertension, liver cirrhosis, HIV infection, and hepatitis virus B or C infection
* History of episodes mimicking demyelinating disorders or a definite diagnosis of multiple sclerosis
* Any creatinine value above 1.5 mg/dl
* Intake of corticosteroids defined as daily intake of prednisone or equivalent more than 1mg/kg for the last three weeks
* Neutropenia defined as <1000 neutrophils/mm3
* Pregnancy or lactation
* History of tuberculosis (latent or active). This will be excluded according to the procedure defined in the screening of patients (see below)
* Major surgery within 28 days prior to Day 0
* It is explicitly stated that intake of antimicrobials for HS is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The efficacy of MABp1 in patients with moderate to severe HS | 12 weeks
  This will be assessed by the difference of achievement of positive HiSCR score between the treatment group and the comparator placebo group at week 12.

SECONDARY OUTCOMES:
The long-term efficacy of MABp1 in patients with moderate to severe HS | Up to 24 weeks
  This will be assessed by the difference of achievement of positive HiSCR score between the treatment group and the comparator placebo group at week 24. Analysis will also be done separately for patients with previous failure or relapse under antiTNF and for patients without previous antiTNF treatment.
The short-and long-term efficacy of MABp1 in the quality of life of patients with moderate to severe HS | Up to 24 weeks
  This will be assessed by the comparisons of dermatology life quality index on all study visits taking also into account the visual analogue scale. Analysis will also be done separately for patients with previous failure or relapse under antiTNF and for patients without previous antiTNF treatment.
The short-and long-term efficacy of MABp1 in individual lesions of patients with moderate to severe HS | Up to 24 weeks
  This will be assessed by the comparisons of modified Sartorius score on all study visits. Analysis will also be done separately for patients with previous failure or relapse under antiTNF and for patients without previous antiTNF treatment.
The effect of MAbp1 on the time to new exacerbation | Up to 24 weeks
  This will be assessed by comparing the time to new exacerbation from week 0 between the two groups of treatment. Analysis will also be done separately for patients with previous failure or relapse under antiTNF and for patients without previous antiTNF treatment.
The effect of MAbp1 on the ultrasonographic findings of the skin lesions | Week 12
  This will be assessed by comparing the changes of skin lesions at week 12 between the two groups of treatment. Analysis will also be done separately for patients with previous failure or relapse under antiTNF and for patients without previous antiTNF treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Institute for the Study of Sepsis; Dimitrios Boumpas, MD, PhD, Principal Investigator — University of Athens
Locations (1):
- 4th Department of Internal Medicine, ATTIKON University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tzanetakou V, Kanni T, Giatrakou S, Katoulis A, Papadavid E, Netea MG, Dinarello CA, van der Meer JWM, Rigopoulos D, Giamarellos-Bourboulis EJ. Safety and Efficacy of Anakinra in Severe Hidradenitis Suppurativa: A Randomized Clinical Trial. JAMA Dermatol. 2016 Jan;152(1):52-59. doi: 10.1001/jamadermatol.2015.3903. PMID 26579854
- [Background] Kimball AB, Jemec GB, Yang M, Kageleiry A, Signorovitch JE, Okun MM, Gu Y, Wang K, Mulani P, Sundaram M. Assessing the validity, responsiveness and meaningfulness of the Hidradenitis Suppurativa Clinical Response (HiSCR) as the clinical endpoint for hidradenitis suppurativa treatment. Br J Dermatol. 2014 Dec;171(6):1434-42. doi: 10.1111/bjd.13270. Epub 2014 Nov 11. PMID 25040429
- [Background] Kanni T, Tzanetakou V, Savva A, Kersten B, Pistiki A, van de Veerdonk FL, Netea MG, van der Meer JW, Giamarellos-Bourboulis EJ. Compartmentalized Cytokine Responses in Hidradenitis Suppurativa. PLoS One. 2015 Jun 19;10(6):e0130522. doi: 10.1371/journal.pone.0130522. eCollection 2015. PMID 26091259
- [Background] Kelekis NL, Efstathopoulos E, Balanika A, Spyridopoulos TN, Pelekanou A, Kanni T, Savva A, Brountzos E, Giamarellos-Bourboulis EJ. Ultrasound aids in diagnosis and severity assessment of hidradenitis suppurativa. Br J Dermatol. 2010 Jun;162(6):1400-2. doi: 10.1111/j.1365-2133.2010.09710.x. Epub 2010 Feb 22. No abstract available. PMID 20184586